CLINICAL TRIAL: NCT02623660
Title: Accelerated Reduction of Post-operative Edema and Early Return to Function Following Total Knee Arthroplasty (TKA)
Brief Title: Microcurrent Stimulation Reduces Post-Operative Swelling and Healing Time Following Knee Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bioelectric Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRC-001
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis of Knee; Edema; Wounds and Injuries
Keywords: Inflammation; Edema; Arthroplasty; Rehabilitation; Replacement; Knee; Total Knee Replacement; Pain, Postoperative; Exercise Therapy; Therapeutics; Early Ambulation; Myofunctional Therapy; Electric Stimulation Therapy; Orthopedic Procedures; Wound Healing; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Edema; Wounds and Injuries; Inflammation; Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): This group will receive treatment from the ODIN1 device in conjunction with standard care and diagnostic device testing.
  Interventions: Device: ODIN1; Other: Standard Care; Device: Diagnostic Device Testing
- Control (Active Comparator): This group will receive the standard care and the diagnostic device testing.
  Interventions: Other: Standard Care; Device: Diagnostic Device Testing

INTERVENTIONS:
Device: ODIN1 — Shortly after surgery, electrodes will be applied to the lower extremity in such a way that the current will flow from the ankle through the knee replacement and pass through the thigh. The frequency of the treatments will vary over the period of time from post-op recovery to end of rehab.
  All treatments are applying current that consists of different combinations of intensities within the micro to nano ampere ranges.
  Arms: Experimental
Other: Standard Care — Anti-thrombotic medication. Elevation and ice. Pain medications as needed. Dressings changes. Topical antibiotics. Progressive physical therapy.
Device: Diagnostic Device Testing — Diagnostic interventions include: the Perometer which scans the lower extremity and determines its volume to a high degree of accuracy; the Impedimed Bioimpedance Spectroscopy (BIS) device that measures intra and intercellular fluid movement; the Microfet muscle force testing device that provides a digital output of the number of pounds exerted by the quadriceps upon extension; the Acumar digital digital Inclinometer that accurately measures the ROM of the knee; and the K.I.S.S. wound measuring system to measure rate of incision healing.

SUMMARY:
The purpose of this study is to determine if patients undergoing a total knee arthroplasty (TKA) experience a clinically significant reduction in healing time when treated post operatively with a specific form of micro and nano-ampere current. The results of this trial will provide a basis for generalizing its outcomes to apply to other joint replacements and revisions by reducing edema and inflammation and therefore will result in a shorter time to heal.

The study will compare electrically treated and non electrically treated patients by using digitally based measurements to determine objective reductions of lower extremity edema including intra and inter cellular shifts in fluid distribution, increased range of motion (ROM) and muscle strength, and improved functional tests of ambulation.

DETAILED DESCRIPTION:
This study is intended to assess the efficiency and efficacy of the ODIN1® microcurrent generating device to reduce post-operative edema, shorten the time to heal and regain maximum function in total knee replacement patients. Changes in swelling will be documented by utilizing a 3D scanning device (Perometer) and a Bio-Impedance Spectroscopy (BIS) device (Impedimed SFB7). These instruments quantitate limb volume and inter and intra-cellular fluid respectively with a high degree of accuracy. Measurements will be made from the first post-operative day until the completion of rehabilitation therapy several months later.

Edema volume and fluid distribution data collected from both control and experimental groups will be compared to determine the statistical significance of the difference between these groups. An additional analysis will be performed on data collected from the non-operated lower limb of each patient.

The second primary objective is to determine the time to complete post-op rehabilitation. Completion will be determined by the ability of the patient to experience an optimal outcome by utilizing performance based measurements of knee function including quadriceps strength and range of motion. The time from surgery to optimal post-op rehabilitation will be recorded.

The determinations of statistical significance between the electrically treated and non-electrically treated groups will be made by analysts on a blind basis. They will not know whether a sample data set is from an experimental or control patient. The codes that document which group the set belongs to will be opened after all analysis is completed by an independent analyst.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be scheduled for a primary total knee replacement surgery
2. Age: 18 - 80 years old
3. Males/Females all ethnicities
4. Must have a minimum serum albumin of 4 and a minimum Hgb of 11
5. Ability to mark appropriately the visual analog scales, keep a log of symptoms, medication use, and ODIN1® use
6. Ability to understand all instructions and the informed consent document before signing it

Exclusion Criteria:

1. Subject younger than 18 years of age
2. Any patient with an electrically implanted device such as a pacemaker, neural stimulator, etc.
3. Subject has any known neoplasms
4. A demonstrated lack of compliance as determined by the Principal Investigator, nurse, or wound care specialist
5. Current participation in another clinical study of an investigational device or drug.
6. Any other condition or finding, which in the opinion of the investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the protocol
7. Subject unwilling or unable to provide informed consent
8. Subjects receiving any medication or having any condition that significantly interferes with the healing process such as a patient taking systemic steroids or immune suppressants or patient has diabetes mellitus with an HbA1c of greater than 7.5, etc.
9. Any female who has experienced menstruation and is less than 5 years postmenopausal shall have a urine pregnancy test before the initial treatment. An additional test will be performed at 3 weeks from the initial treatment date. Any subject with a positive pregnancy test shall be excluded
10. Subjects with significant peripheral extremity lymph edema
11. Subjects with Stage III or IV peripheral vascular disease, as defined by the Fontaine stages
12. Subjects with venous insufficiencies of Class III or greater, as defined by the Comprehensive Classification System for Chronic Venous Disorders (CEAP)
13. Subjects with muscle skeletal disorders that are not related to the knee
14. Subjects with uncontrolled Blood Pressure
15. Subjects with neurological disease affecting locomotion
16. Subjects with BMI > 35
17. Subjects that are active smokers
18. Subjects that live on the second floor or higher without elevator access
19. Subjects must not have had a prior TKA. This study is for Primary TKA patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Reduction of post-operative edema | 120 days
  Determine the rate of reduction in edema by measuring the volume changes in the operated lower extremity over time
Decrease in time to heal | 120 Days
  Determine the rate of healing by measuring the time elapsed from surgery to reach optimal function by measuring muscle strength, range of knee motion, standardized rehabilitation testing designed to quantitatively measure ambulation. When these measurements show no signs of improvement for a period of 30 days or greater, then the time elapsed after surgery until the beginning of this 30 day or greater period will be recorded and used as a measure of time to heal.

SECONDARY OUTCOMES:
Reduction of pain | 90 days
  Record the degree of pain experienced by measuring the pain level on the universal pain scale of 1-10 over time elapsed since surgery.
Reduction of bacterial infections | 60 Days
  Compare the incidence of TKA related infections in all participants. The measurement will be the number of recorded infections, related to the surgery, that has occurred within the first 60 days of that surgery in all participants. That number will be compared between the experimental and the control groups.
Increased healing of the surgical incision | From the 1st post-op day until 60 Days post-op
  Photograph and rate incision healing from 1st post-op day through day 60 comparing all participants.
Reduction of Pain Medication Usage | 90 days
  Record the consumption of all pain medications consumed to mitigate post-operative pain. A total dosage will be calculated in terms of morphine equivalent strengths and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Hillock, M.D., Principal Investigator — Centennial Hills Hospital & University of Nevada School of Medicine
Locations (2):
- United States (2):
  - Nevada Orthopedic and Spine Center, Las Vegas, Nevada
  - Centennial Hills Hospital, Las Vegas, Nevada

REFERENCES:
- [Background] Shi R, Borgens RB. Three-dimensional gradients of voltage during development of the nervous system as invisible coordinates for the establishment of embryonic pattern. Dev Dyn. 1995 Feb;202(2):101-14. doi: 10.1002/aja.1002020202. PMID 7734729
- [Background] Hotary KB, Robinson KR. Endogenous electrical currents and voltage gradients in Xenopus embryos and the consequences of their disruption. Dev Biol. 1994 Dec;166(2):789-800. doi: 10.1006/dbio.1994.1357. PMID 7813796
- [Background] Soong HK, Parkinson WC, Bafna S, Sulik GL, Huang SC. Movements of cultured corneal epithelial cells and stromal fibroblasts in electric fields. Invest Ophthalmol Vis Sci. 1990 Nov;31(11):2278-82. PMID 2242993
- [Background] Zhao M, Dick A, Forrester JV, McCaig CD. Electric field-directed cell motility involves up-regulated expression and asymmetric redistribution of the epidermal growth factor receptors and is enhanced by fibronectin and laminin. Mol Biol Cell. 1999 Apr;10(4):1259-76. doi: 10.1091/mbc.10.4.1259. PMID 10198071
- [Background] Lin F, Baldessari F, Gyenge CC, Sato T, Chambers RD, Santiago JG, Butcher EC. Lymphocyte electrotaxis in vitro and in vivo. J Immunol. 2008 Aug 15;181(4):2465-71. doi: 10.4049/jimmunol.181.4.2465. PMID 18684937
- [Background] McCaig CD, Rajnicek AM, Song B, Zhao M. Controlling cell behavior electrically: current views and future potential. Physiol Rev. 2005 Jul;85(3):943-78. doi: 10.1152/physrev.00020.2004. PMID 15987799
- [Background] Sato MJ, Kuwayama H, van Egmond WN, Takayama AL, Takagi H, van Haastert PJ, Yanagida T, Ueda M. Switching direction in electric-signal-induced cell migration by cyclic guanosine monophosphate and phosphatidylinositol signaling. Proc Natl Acad Sci U S A. 2009 Apr 21;106(16):6667-72. doi: 10.1073/pnas.0809974106. Epub 2009 Apr 3. PMID 19346484
- [Background] Li L, Gu W, Du J, Reid B, Deng X, Liu Z, Zong Z, Wang H, Yao B, Yang C, Yan J, Zeng L, Chalmers L, Zhao M, Jiang J. Electric fields guide migration of epidermal stem cells and promote skin wound healing. Wound Repair Regen. 2012 Nov-Dec;20(6):840-51. doi: 10.1111/j.1524-475X.2012.00829.x. Epub 2012 Oct 19. PMID 23082865
- [Background] Man IO, Markland KL, Morrissey MC. The validity and reliability of the Perometer in evaluating human knee volume. Clin Physiol Funct Imaging. 2004 Nov;24(6):352-8. doi: 10.1111/j.1475-097X.2004.00577.x. PMID 15522044
- [Background] Pichonnaz C, Bassin JP, Currat D, Martin E, Jolles BM. Bioimpedance for oedema evaluation after total knee arthroplasty. Physiother Res Int. 2013 Sep;18(3):140-7. doi: 10.1002/pri.1540. Epub 2012 Nov 27. PMID 23188719